CLINICAL TRIAL: NCT05776004
Title: A Randomized, Double-Blind, Placebo-Controlled Multicenter Study to Evaluate the Efficacy and Safety of CAL02 Administered Intravenously in Addition to Standard of Care in Subjects With Severe Community-Acquired Bacterial Pneumonia (SCABP)
Brief Title: Blinded Efficacy and Safety Study of CAL02 IV Plus SOC in Subjects With Severe Community-Acquired Bacterial Pneumonia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Eagle Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EGL-6535-C-2202
Record Dates: First submitted 2023-02-14; First posted 2023-03-20 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Pneumonia, Bacterial
Keywords: Community-Acquired
MeSH Terms: conditions — Pneumonia, Bacterial

STUDY DESIGN:
Intervention Model Description: Adaptive, randomized, double-blind, placebo-controlled study
Who Masked: Participant, Investigator
Masking Description: Placebo-controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CAL02 with Standard of Care (Experimental): CAL02 (a mixture of 2 liposomal components, both empty, unilamellar, liposomes) will be administered as 2, IV infusions, 24 - 26 hours apart in addition to Standard of Care therapy for SCABP, according to scientific guidelines. CAL02 infusions will be administered over a 1 -2 hour period.
  Interventions: Drug: CAL02
- Placebo (Placebo Comparator): Placebo will be administered as 2, IV infusions, 24 - 26 hours apart in addition to Standard of Care therapy for SCABP, according to scientific guidelines. Placebo will be prepared and administered following the same infusion protocol as CAL02. Placebo infusions will be administered over a 1 to 2 hour period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CAL02 — CAL02 consists of a mixture of 2 liposomes and is a non-biological bacterial virulence neutralizer.
  Arms: CAL02 with Standard of Care
Drug: Placebo — Physiological 0.9% sodium chloride solution for iv administration
  Arms: Placebo

SUMMARY:
This is a placebo-controlled study to evaluate the addition of CAL02 to standard of care in treating hospitalized subjects diagnosed with severe community acquired bacterial pneumonia (SCABP) requiring critical care measures

DETAILED DESCRIPTION:
Subjects diagnosed with SCABP and requiring critical care measures, will receive either 2 intravenous infusions of CAL02 (13.7 to 24 mg/kg bracketed dose by weight), administered 24-26 hours apart or 2 intravenous infusions of placebo. Additionally, all subjects will receive standard of care (SOC) therapy for SCABP, according to scientific guidelines. Critical care measures provide intensive and specialized medical and nursing care, a capacity for continuous monitoring 24 hours/day, and multiple modalities of physiologic organ support to sustain life in seriously/critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* male or females older than 18 years old
* Body Weight 40 - 140 kg;
* clinical diagnosis of CABP diagnosed less than or equal to 48 hrs after hospital admission;
* presence of at least one of the protocol defined SCABP severity criteria:
* at least two clinical symptoms
* at least 2 vital sign abnormalities
* at least one finding of other clinical signs/laboratory abnormalities
* radiographic evidence in support of pneumonia with likely bacterial origin
* presence of at least one of the following severity criteria based on protocol defined SCABP:
* respiratory failure requiring invasive mechanical ventilation support
* respiratory failure requiring non-invasive positive pressure ventilation support
* respiratory failure requiring high-flow oxygen
* septic shock requiring treatment with vasopressors at therapeutic doses for at least 2 hours
* requires critical care for management of SCABP
* onset of severity criteria less than 48 hours from diagnosis of CABP or upon discussion with medical monitor
* written informed consent before any study-specific assessment is performed

Exclusion Criteria: Subjects in the hospital who meet any of the following criteria at screening and before study drug administration:

* subjects with ventilator-associated pneumonia, aspiration pneumonia, fungal pneumonia, viral pneumonia (viral coinfection may be exempted subject to discussion with medical monitor);
* subjects more than 12 hours from the diagnosis of SCABP;
* SOFA score greater than 12 points
* subject received IV antibiotics for CABP/SCABP for more than 48 hours at the time of randomization if sensitivity supports appropriate empiric therapy chosen and administered
* renal replacement therapy
* known hypersensitivity to liposomal formulations
* end-stage neuromuscular disorders, tracheostomy, known bronchial obstruction, post-operative aspiration pneumonia, cystic fibrosis, known or suspected pneumocystis jirovecii or tuberculosis pneumonia, post organ transplant, or primary or metastatic malignancy in the lungs
* current or recent participation in an investigational study (within 30 days of screening or 5 half-lives of the investigational compound, whichever is longer)
* known liver dysfunction, chronic liver disease with Child Pugh C or esophageal varices
* moribund clinical conditions at the time of screening or time of the first study medication infusion
* refractory septic shock at the time of randomization
* subject has any medical disease or condition that, in the opinion of the investigator, compromises the subject's safety or compromises the interpretation of results
* nursing and pregnant women
* women of childbearing potential and non-surgically sterile males

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Estimated)
Dates: Start 2023-07-22 (Actual); Primary Completion 2026-02-10 (Estimated); Study Completion 2026-09-07 (Estimated)

PRIMARY OUTCOMES:
Efficacy- clinical recovery | 28 days
  To evaluate the effect of CAL02 administration on clinical recovery compared to placebo. The time (days) to clinical recovery will be measured, as defined by the day all disease severity criteria which led to SCABP diagnosis per protocol at randomization and any new severity criteria which occurred after randomization are resolved, and no repeat or additional severity criteria are met within 24 hours after clinical recovery.
Incidence of Treatment-Emergent Adverse Events | 28 days
  To evaluate the safety and tolerability of CAL02 versus placebo. The number of participants with treatment-emergent adverse events including IV infusion-related reactions, and the number of participants with study drug dosing interruptions and discontinuations will be measured.

SECONDARY OUTCOMES:
Critical Care Management | 28 days
  To evaluate the effect of CAL02 administration on the duration of critical care management compared to placebo. The time (days) participant remains in hospital critical care from randomization until discharge will be measured.
Hospital Stay | 28 days
  To evaluate the effect of CAL02 administration on the duration of overall hospital stay compared to placebo. The time (days) participant remains in hospital from randomization until discharge will be measured.
Early Clinical Recovery | 5 days
  To evaluate the effect of CAL02 administration on early clinical recovery (by Day 5) compared to placebo. The number of participants who achieve clinical recovery by Day 5 will be assessed; clinical recovery as defined by the day all disease severity criteria which led to SCABP diagnosis per protocol at randomization and any new severity criteria which occurred after randomization are resolved, and no repeat or additional severity criteria are met within 24 hours after clinical recovery.
Organ Failure Assessment Scores | 7 days
  To evaluate the effects of CAL02 administration on Sequential Organ Failure Assessment (SOFA) scores compared to placebo. The minimum total score is 0 and the maximum total score is 24. A higher total SOFA score indicates worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Valentin R Curt, MD, Study Chair — Eagle Pharmaceuticals, Inc.
Locations (90):
- United States (7):
  - UCSF Hospital, Fresno, California
  - UF Health Shands Hospital, Gainesville, Florida
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Wake Forest Baptist Health Hospital, Winston-Salem, North Carolina
  - Cleveland Clinic Fairview Hospital, Cleveland, Ohio
  - University of Texas Medical Branch, Galveston, Texas
- Argentina (4):
  - Hospital Interzonal General de Agudo Dr Jose Pena, Bahía Blanca, Buenos Aires
  - Hospital Italiano de Buenos Aires, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Hospital Misericordia Nuevo Siglo, Córdoba
  - Hospital Central, Mendoza
- Belgium (3):
  - Clinique Universitaire Saint Luc, Brussels
  - Clinique Saint Pierre, Ottignies
  - Chu-Ucl-Namur, Yvoir
- Brazil (4):
  - Hospital Mae de Deus, Porto Alegre, Rio Grande do Sul
  - Fundacao Faculdade Regional de Medicina de Sao Jose do Rio Preto, São José do Rio Preto, São Paulo
  - Unidade de Pesquisa Clinica da Faculdade de Medicina de Botucatu, Botucatu
  - Hospital do Servidor Publico Estadual, São Paulo
- Canada (5):
  - Foothills Hospital Medical Centre, Calgary, Alberta
  - Peter Lougheed Centre, Calgary, Alberta
  - Rockyview General Hospital, Calgary, Alberta
  - South Health Campus Hospital, Calgary, Alberta
  - Saint Paul's Hospital, Vancouver
- Pontificia Universidad Catolica de Chile, Santiago, Chile
- Colombia (2):
  - Centro de Investigacion Clinica de la Costa SAS, Barranquilla
  - Fundacion Cardioinfantil - Instituto de Cardiologia, Bogotá
- Czechia (3):
  - Krajska Zdravotni, a.s., Teplice
  - Krajska Zdravotni, a.s., Ústí nad Labem
  - Oblastní nemocnice Kolín, a.s., nemocnice Středočeského kraje, Zizkova
- France (14):
  - CHD Vendee, La Roche-sur-Yon, Vendee
  - CHU Angers, Angers
  - Centre Hospitalier Victor Dupouy, Argenteuil
  - Hopital Nord Franche Comte, Belfort
  - Hospital Fleyriat, Bourg-en-Bresse
  - Centre Hospitalier de Dieppe, Dieppe
  - Plateforme de Biologie Hospitalo-Universitaire, Dijon
  - Hopital Raymond Poincare, Garches
  - Pole Urgences Medecine Aigue CHU de Grenoble-Alpes, Grenoble
  - Hospital Dupuytren, Limoges
  - Centre Hospitalier de Melun-Senart, Melun
  - CHU de Nantes, Nantes
  - Hopitaux Universitaires de Strasbourg - Nouvel Hopital Civil, Strasbourg
  - Centre Hospitalier Bretagne Atlantique, Vannes
- Georgia (7):
  - LTD Batumi Medical Center, Batumi
  - JSC Rustavi Central Hospital, Rustavi
  - LLC Aleksandre Aladashvili Clinic, Tbilisi
  - LTD Tbilisi Central Hospital, Tbilisi
  - LTD Simon Khechinashvili University Hospital, Tbilisi
  - The First Medical Center LTD, Tbilisi
  - LTD N5 Clinical Hospital, Tbilisi
- Greece (3):
  - Thoracic General Hospital, Athens
  - University General Hospital Attikon, Athens
  - University General Hospital, Heraklion
- Hungary (4):
  - Bekes Varmegyei Kozponti K6rhaz, Gyula
  - Szaboles-Szatmar-Bereg Varmegyei Oktatokorhaz, Nyíregyháza
  - Borsod-Abauj-Zemplen Varmegyei Kozponti Korhaz es Egyetemi Oktatov, Szentpeteri Kapu
  - Zala Varmegyei Szent Rafael Korbaz, Zalaegerszeg
- Latvia (3):
  - Liepajas Regional Hospital, Liepāja
  - Pauls Stradins Clinical University Hospital, Riga
  - Vidzemes Hospital, Valmiera
- Peru (5):
  - Hospital Nacional III, Arequipa
  - Clinica Ricardo Palma, Lima
  - Clinica San Pablo-Sede Surco, Lima
  - Hospital Nacional Edgardo Rebagliati, Lima
  - Hospital de la Amistad, Piura
- Romania (5):
  - Pius Brinzeu County Emergency Clinical Hospital, Timișoara, Judet Timis
  - Elias University Emergency Hospital, Bucharest
  - Fundeni Clinical Institute, Bucharest
  - Cluj County Emergency Clinical Hospital, Cluj-Napoca
  - Bihor County Emergency Clinical Hospital, Oradea
- Serbia (4):
  - University Clinical Centre of Serbia, Belgrade
  - Institute for Pulmonary Diseases, Kamenitz
  - University Clinical Centre, Kragujevac
  - University Clinical Centre, Niš
- Univerzitna nemocnica, Martin, Slovakia
- South Africa (5):
  - Helen Joseph Academic Hospital, Johannesburg, Gauteng
  - FCRN Clinical Trial Centre, Vereeniging, Gauteng
  - Tygerberg Hospital, Cape Town
  - Ryexo Clinical Research, Pretoria
  - Dr JM Engelbrecht Trial Site, Somerset West
- Spain (10):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Parc Tauli Hospital Universitari, Barcelona
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario Infanta Leonor, Madrid
  - C.H.U de Santiago de Compostela, Santiago de Compostela
  - Hospital Universitario de Tarragona Joan XXIII, Tarragona
  - Hospital Universitari Mutua Terrassa, Terrassa
  - Hospital Universitario de Toledo, Toledo
  - Hospital Universitario Dr Peset, Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid